CLINICAL TRIAL: NCT04761679
Title: Nasal Bridge Pressure Injury Prevention Using Protective Dressing and Halyard Fluidshield N95 Mask
Brief Title: Nasal Bridge Pressure Injury Prevention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Evolution of the COVID19 pandemic with subsequent spread to all areas of clinical care severely affected the number of potential participants that were able to safely participate in the study.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT2889
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Pressure Ulcer of Skin; Pressure Injury
Keywords: Pressure Injury Prevention; Personal Protective Equipment; Nursing; Nasal Bridge; N-95 Mask
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Applying the Mepilex foam
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Applying the Mepilex foam — Mepilex foam will be directly applied on the nasal bridge directly between the skin and the N95 mask.
  Arms: Intervention Group

SUMMARY:
The primary goal of this study is to explore whether applying the Mepilex foam on the nasal bridge directly between the skin and the N95 mask will prevent nasal bridge pressure injury among nursing staff, secondary to long-term ( >8+ hours) wear time. The secondary goal is to evaluate if using the Mepilex maintains the seal of the mask.

DETAILED DESCRIPTION:
Nurses use the N95 Mask as part of the personal protective equipment (PPE) when caring for patients with COVID-19. The N95 mask covers their nose and mouth with a tight seal. Nurses wear the mask for more than 8 hours per day, as a result they are at increased risk for skin injury on the nasal bridge. Mepliex is foam dressing which has been used to prevent pressure injuries to the skin. This study will evaluate if using Mepilex or band-aid on the nasal bridge of the nurses who wear the N95 for more than 8 hours decreases the potential for skin injury. In addition, the investigators will test if the Mepilex or band-aid also maintains the seal of the mask. Maintaining the seal is important to ensure that the nurse is not exposed to the virus. The investigators will be working with nurses who do not directly take care of COVID-19 patients to ensure the safety of all participants.

ELIGIBILITY:
Inclusion Criteria:

* The sample will consist of nursing staff working on non-COVID units, including: Medical Surgical Units, Operating Rooms or Ambulatory Care- Labor and Delivery Unit, Maternity Unit and Medical Oncology Unit, at NewYork-Presbyterian (NYP) Lawrence Hospital.

Exclusion Criteria:

* Exclusion Criteria: A score on > 5 the COVID Anxiety Scale. The scale has 4 questions with 5 possible options (rated 1 - 5), to evaluate the effect of COVID19 on the individual. The lowest possible score is 0, the highest possible score is 20. A score of 5 states that the individual experiences COVID19 related anxiety for 'Rarely' or 'Not at All". Excluding participants with a score of > 5 will prevent unnecessary harm to study participants or exacerbate symptoms of anxiety.
* Nurses working in the Emergency Department, Intensive Care Unit or a unit with a focus on the exposed COVID-19 population
* Non-clinical nurses, volunteer or agency registered nurses
* Known history of skin breakdown or damage to the nasal bridge
* History of skin-related conditions including (acne vulgaris, Psoriasis, Herpetic lesions to mouth, nasal areas)
* History of surgery to nasal bridge
* Pregnant nurses in their third trimester
* History of respiratory extended respirator use in addition to the hours collected in this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Pressure Injury Prevention | 48 hours
  Researchers will count the number of participants with and without injury on the nasal bridge directly between the skin and the N95 mask

SECONDARY OUTCOMES:
Number of Participants that Maintain Mask Seal Integrity | 12 hours
  Researchers will assess the integrity of the N95 mask seal using both interventions - Mepilex and Band-Aid. The number of participants with acceptable seal according to the Fit Test will be counted

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Holder, MSN, RN, ACCNS-AG, CCRN, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded participant data will be made available to future researchers with a goal to replicate this study and add to the body of nursing knowledge